CLINICAL TRIAL: NCT05678205
Title: A Multicenter, Open-label, Phase 1/2 Clinical Trial to Evaluate the Safety and Anti-Tumor Activity of AB-201 in Subjects With Advanced HER2+ Solid Tumors
Brief Title: A Clinical Trial of the Safety and Anti-Tumor Activity of AB-201 in Subjects With Advanced HER2+ Solid Tumors
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Corporate business decision
Sponsor: Artiva Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AB-201-01
Record Dates: First submitted 2022-12-23; First posted 2023-01-10 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Gastric Cancer; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Phase 1 Dose Confirmation (Experimental): Dose Confirmation of AB-201 in advanced metastatic breast cancer, gastric or gastroesophageal junction adenocarcinoma with HER2 overexpression
  Interventions: Drug: AB-201; Drug: Cyclophosphamide; Drug: Fludarabine
- Phase 2 Cohort A (Experimental): AB-201 given to patients with advanced/unresectable or metastatic breast cancer with HER2 overexpression (IHC ≥2+) that is refractory to or intolerant of standard treatment, or for which no standard treatment is available
  Interventions: Drug: AB-201; Drug: Cyclophosphamide; Drug: Fludarabine
- Phase 2 Cohort B (Experimental): AB-201 given to patients with advanced/unresectable or metastatic breast cancer with HER2 overexpression (IHC 3+ or IHC 2+/ISH+) that is relapsed to, refractory to, or intolerant of previous trastuzumab deruxtecan (T-DXd) based therapy
  Interventions: Drug: AB-201; Drug: Cyclophosphamide; Drug: Fludarabine
- Phase 2 Cohort C (Experimental): AB-201 given to patients with advanced/unresectable or metastatic gastric or gastroesophageal junction adenocarcinoma with HER2 overexpression (IHC ≥ 2+) that is refractory to or intolerant of standard treatment, or for which no standard treatment is available
  Interventions: Drug: AB-201; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: AB-201 — NK Cell Therapy
Drug: Cyclophosphamide — Lymphodepleting chemotherapy
Drug: Fludarabine — Lymphodepleting chemotherapy

SUMMARY:
This clinical trial will enroll subjects with HER2+ solid tumors and is conducted in two phases. The primary objective of Phase 1 is to determine the safety and tolerability of AB-201 in subjects with advanced HER2+ solid tumors. The primary objective of Phase 2 is to evaluate the efficacy of AB-201.

Subjects will receive up to 3 doses of AB-201, followed by scheduled assessments of overall health and tumor response.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status 0 to 1.
* Histologically confirmed HER2 expressed breast or gastric/GEJ cancer IHC ≥ 2+ within 6 months prior to study entry.
* Confirmed diagnosis of an advanced/unresectable or metastatic HER2+ breast or gastric/GEJ cancer that is refractory to, or intolerable of standard treatment, or for which no standard treatment is available.
* Must have received prior cancer therapy: Subjects with breast cancer must have received ≥ 2 prior systemic therapies; subjects with gastric/GEJ cancer must have received ≥ 1 prior systemic therapy(ies); subjects with IHC 3+ or IHC 2+/ISH+ cancers must have received previous treatment with a HER2-targeting therapy.

Exclusion Criteria:

* Known past or current malignancy other than inclusion diagnosis.
* Known clinically significant cardiac disease.
* Active central nervous system (CNS) metastases, or involvement of the CNS, unless there is a history of at least 3 months of sustained remission.
* Unresolved toxicities from prior anticancer therapy.
* Ongoing uncontrolled systemic infections requiring antibiotic, anti-fungal, or anti-viral therapy.
* History of sensitivity or intolerance to cyclophosphamide or fludarabine.
* Pregnant or lactating females and subjects of both sexes who are not willing to practice birth control from the time of consent through 6 months after administration of the last AB-201 dose.
* Severe disease progression or health deterioration within 2 weeks prior to lymphodepletion regimen.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Safety: incidence and severity of adverse events and serious adverse events | From the time of consent through End of Study (up to 18 months per patient)
Determination of Recommended Phase 2 Dose (RP2D): safety, preliminary efficacy (based on objective response rate (ORR) defined as the proportion of patients with a complete or partial response) and pharmacokinetics | From the time of consent through End of Study (up to 18 months per patient)
Efficacy: Objective Response Rate, defined as the proportion of patients with a complete or partial response | From the time of consent through End of Study (up to 18 months per patient)

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Graef, MD, Ph.D, Study Director — Artiva Biotherapeutics
Locations (2):
- Oregon Health Science University (OHSU), Portland, Oregon, United States
- The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No